CLINICAL TRIAL: NCT06313944
Title: German (GE) Multicenter Prospective Data Collection (Registry) on Treatment With Transcranial Pulse Wave Stimulation (TPS) in Patients With Alzheimer's Disease (A)
Brief Title: German Registry of Alzheimer's Disease Treated With Transcranial Pulse Stimulation
Acronym: GE-R-A-TPS
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Storz Medical AG (Industry)
Responsible Party: Sponsor
Other Study IDs: GE-R-A-TPS
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Transcranial Pulse Wave Stimulation (TPS)
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Clinical Alzheimer's syndrome treated with TPS: Patients with clinical Alzheimer's syndrome, defined by a gradually progressive change in memory function (for severity using the MMSE as a screening tool) and impairment of activities of daily living for more than six months that have planned treatment with TPS
  Interventions: Diagnostic Test: Registry

INTERVENTIONS:
Diagnostic Test: Registry — Clinical data collection of patients scheduled for on-label treatment

SUMMARY:
This study will primarily investigate the safety and secondarily the effect and applicability of Transcranial Pulse Wave Stimulation (TPS) for the treatment of Alzheimer's disease in the context of a PMCF study (Post-Market Clinical Follow-up). The multicenter, prospective data collection should help to optimize the stimulation protocol, as well as to record frequent to occasional adverse effects of the product and cognitive, affective and subjective scores.

DETAILED DESCRIPTION:
This study will primarily investigate the safety and secondarily the effect and applicability of Transcranial Pulse Wave Stimulation (TPS) for the treatment of Alzheimer's disease in the context of a PMCF study (Post-Market Clinical Follow-up). The multicenter, prospective data collection should help to optimize the stimulation protocol, as well as to record frequent to occasional adverse effects of the product and cognitive, affective and subjective scores. Adverse effects and adverse events without a clear causal relationship will be documented in terms of frequency and severity. Furthermore, the progression of improvement in Alzheimer's symptoms as a result of TPS treatment is summarized in various neuropsychological scales.

ELIGIBILITY:
Inclusion Criteria:

i. Age = 18 to 85 ii. N>=100, clinical Alzheimer's syndrome, defined by a gradually progressive change in memory function (for severity using the MMSE as a screening tool) and impairment of activities of daily living for more than six months iii. MRI scan, in vivo evidence from CSF and/or PET using the NIA-AA criteria, which categorize the underlying pathological processes based on biomarkers, should be added if possible, but are optional. These biomarkers are categorized as ß-amyloid deposition, pathological tau and neurodegeneration [AT(N)], which can be detected on imaging and in biofluids. If possible, patients with Alzheimer's disease (AD) or Alzheimer's continuum should be included.

iv. TPS treatment in a center of a neurological or psychiatric specialist and performed under supervision of a specialist

Exclusion Criteria:

i. Relevant intracerebral pathologies not related to Alzheimer's disease, such as vascular encephalopathy Fazekas grade 3, tumors, vascular malformations, pregnancy, metal implants, CAA according to Boston criteria, Z.n. or during antibody therapy ii. Blood coagulation disorders or oral anticoagulation iii. Epilepsy iv. Medical conditions leading to non-compliance with the protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AD Patients undergoing TPS
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of (Serious) Adverse Events | through study completion, an average of 1 year
  Number of adverse events (without causal relationship to therapy) AE, SAE (query after the first 6-cycle block and before each booster) scaling according to NRS (1-10) for each ADE (query before each stimulation)
Number of adverse device effects | through study completion, an average of 1 year
  Number of ADEs and (U)SADEs scaling according to NRS (1-10) for each ADE (query before each stimulation)

SECONDARY OUTCOMES:
ADAS | Baseline, post first 6 sessions and after 3, 6, 9 and 12 months
  Alzheimer's Disease Asessment Scale (ADAS) baseline and post 6 sessions as well as after 3, 6, 9 and 12 months (desired but not mandatory, collected within 3 days after stimulation)
Mini Mental State Examination (MMSE) baseline and follow- up | Baseline, post first 6 sessions and after 3, 6, 9 and 12 months
  Mini Mental State Examination (MMSE) baseline and post 6 sessions as well as after 3, 6, 9 and 12 months (desired but not mandatory, collected within 3 days after stimulation)
BDI-II | Baseline, post first 6 sessions and after 3, 6, 9 and 12 months
  BDI-II baseline and post 6 sessions as well as after 3, 6, 9 and 12 months (desired but not mandatory, collected within 3 days after stimulation)
Clinical Dementia Rating Sum of Boxes Score (CDR-SB) | Baseline, post first 6 sessions and after 3, 6, 9 and 12 months
  Clinical Dementia Rating Sum of Boxes Score (CDR-SB) baseline and post 6 sessions as well as after 3, 6, 9 and 12 months (desired but not mandatory, collected within 3 days after stimulation)
Alzheimer's Disease Cooperative Study/ Activities of Daily Living Scale (ADCS-ADL) | Baseline, post first 6 sessions and after 3, 6, 9 and 12 months
  Alzheimer's Disease Cooperative Study/ Activities of Daily Living Scale (ADCS-ADL) at baseline and post 6 sessions as well as after 3, 6, 9 and 12 months (desired but not mandatory, collected within 3 days after stimulation)

OTHER OUTCOMES:
Numeric Rating Scale (NRS) for the main symptom | 12 months
  Numeric Rating Scale (NRS) for the main symptom

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wojtecki, Prof. Dr., Principal Investigator — Heinrich-Heine-Universität
Locations (4):
- Germany (4):
  - Ernst von Bergmann Klinikum - Klinik für Neurologie und Klinische Neuropsychologie, Potsdam, Brandenburg
  - Universitätsklinikum Bonn - Klinik für Parkinson, Schlaf- und Bewegungsstörungen, Bonn, North Rhine-Westphalia
  - Hospital zum Heiligen Geist GmbH & Co KG Klinik für Neurologie und Neurorehabilitation, Kempen
  - Praxis Dr. Schwarz, Ulm